CLINICAL TRIAL: NCT02312102
Title: Phase I Dose Escalation Study of Velcade in Combination With Lenalidomide in Patients With Relapsed Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) After Allogeneic Stem Cell Transplantation
Brief Title: Velcade and Lenalidomide in Patients With Relapsed AML and MDS After Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celgene Corporation (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew Mark Brunner, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-213
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: myelodysplastic syndrome; acute myeloid leukemia; allogeneic stem cell transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade and Lenalidomide (Experimental): Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  Each treatment cycle lasts 28 days (4 weeks). The first two cycles are called the induction cycles. If the participant respond to treatment during the first two cycles, they can continue on to the maintenance cycles.
  During the induction and maintenance cycles, patients receive up to the MTD of lenalidomide on days 1-21 days only. During days 22-28 (4th week) there is a rest period.
  Bortezomib: During the induction cycles, the medication will be given on days 2, 5, 9, and 12 followed by a 17-day rest period. During the maintenance cycles, bortezomib will be given on days 2, and 5 followed by 23-day rest period.
  Interventions: Drug: Lenalidomide; Drug: Velcade

INTERVENTIONS:
Drug: Lenalidomide — Chemotherapy
  Other Names: Revlimid
Drug: Velcade — Chemotherapy
  Other Names: bortezomib

SUMMARY:
This research study is evaluating drugs called bortezomib and lenalidomide as a possible treatment for myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

The purpose of this research study is to determine the safety and efficacy of the bortezomib and lenalidomide investigational combination. This drug combination has been used in the treatment of relapsed/refractory multiple myeloma and has been previously investigated in the treatment of MDS and AML, albeit at a lower dose of lenalidomide. In this research study, the investigators are looking for the highest dose of the combination that can be given safely and see how well it works as a combination for MDS and AML in individuals whose disease has relapsed after an SCT.

DETAILED DESCRIPTION:
* After the screening procedures confirm participation in the research study:
* The participant will be given a study drug-dosing calendar for each treatment cycle. The investigators are looking for the highest dose of the combination of study drugs that can be administered safely without severe or unmanageable side effects in participants that have, not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.
* Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
* Each treatment cycle lasts 28 days (4 weeks). The first two cycles are called the induction cycles. If the participant respond to treatment during the first two cycles, they can continue on to the maintenance cycles.

  * Lenalidomide
  * Bortezomib:

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* A diagnosis of recurrent, persistent, or progressive acute myelogenous leukemia (AML), defined as >= 5% blasts in a patient with known prior history of AML, or recurrent, persistent, or progressive myelodysplastic syndrome (MDS) according to WHO criteria.
* Must have undergone an allogeneic SCT (regardless of stem cell source)
* Patients must be 18 years or older
* Able to adhere to study schedule and other protocol requirements
* Must be off all immunosuppressive medications (except prednisone) for at least 2 weeks prior to study entry.
* Must be on less than 21 mg of oral prednisone daily for GVHD
* ECOG performance status 0-2 (see Appendix 2)
* Participants must have the following organ function all within 21 days prior to enrollment

  * Total bilirubin ≤ 2.0 mg/dl unless due to underlying conjugation disease such as Gilbert's
  * ALT and AST ≤ 3X the upper limit of normal
  * Creatinine < 2.0 mg/dl
* Patients may receive hydroxyurea or leukopheresis as necessary
* Patients must give voluntary written informed consent and HIPA authorization before performance of any study-related procedure not part of normal medical care with the understanding that consent maybe withdrawn by the subject at any time without prejudice to future medical care.
* All previous cancer therapy including donor lymphocyte infusions must have been discontinued at least 2 weeks prior to treatment in this study.
* All study participants must be registered in the RevREMS® program and be willing and able to comply with the requirements of REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Ejection fraction < 40% obtained by either MUGA or echocardiogram
* Patients who had had a myocardial infarction within 6 months of enrollment or have New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the consent form.
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at an unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patients with major surgery within 28 days prior to trial enrollment
* Patients with greater than or equal to grade 2 peripheral neuropathy or active herpes infection
* Patients with ≥ grade 3 acute graft-versus-host disease are excluded from the study
* Patients with moderate or severe chronic graft-versus host requiring more than 20 mg of oral prednisone therapy are excluded from the study.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cirrhosis, chronic obstructive or restrictive pulmonary disease, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Patients with any serious or medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Female subject is pregnant or breast-feeding. Lactating females must agree not to breastfeed while taking lenalidomide.
* Patient has received an investigational drug within 14 days of enrollment
* Known hypersensitivity to thalidomide or lenalidomide
* Known hypersensitivity to Velcade, boron, or mannitol
* The development of erythema nodosum as characterized by desquamating rash while taking thalidomide or similar drugs
* Concurrent use of other anti-cancer agents or treatment
* Known positive for HIV
* Diagnosed or treated for a non-hematologic malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
MTD of Bortezomib and Lenalidomide, | 28 days
  Maximum tolerated dose

SECONDARY OUTCOMES:
Assess clinical efficacy in terms of the number of patients experiencing a decrease in blast percentage. | 2 Years
  Change in blasts during treatment
Document the remission frequency in patients receiving up to 2 induction cycles of high-dose lenalidomide combined with Velcade. | Day 42
  Remission rate
Percentage of Complete Response | Baseline, Day 84
  Overall response rate
Percentage of Participants with Disease Free Survival( DFS ) | 2 Years
  Disease free survival
Percentage of Overall Survival | 2 Years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Brunner, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided